CLINICAL TRIAL: NCT00910780
Title: Metabolic Effects of Antipsychotic Substitution in Children
Acronym: SMEAC
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Study was not funded.
Sponsor: Washington University School of Medicine (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-0858
Record Dates: First submitted 2009-05-28; First posted 2009-06-01 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-03

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Aripiprazole; Olanzapine; Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Staying on Risperdal (Active Comparator)
  Interventions: Drug: Risperdal
- Risperdal switched to Abilify (Active Comparator)
  Interventions: Drug: Aripiprazole
- Staying on Zyprexa (Active Comparator)
  Interventions: Drug: Zyprexa
- Zyprexa switched to Abilify (Active Comparator)
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole — via oral tablets, everyday
  Arms: Risperdal switched to Abilify; Zyprexa switched to Abilify
Drug: Zyprexa — via oral tablets, taken once daily
  Arms: Staying on Zyprexa
Drug: Risperdal — via oral tablets, taken once daily
  Arms: Staying on Risperdal

SUMMARY:
This project aims to identify whether therapeutic substitution of aripiprazole for risperidone or olanzapine, combined with standard nutrition intervention, will impact the metabolic changes associated with antipsychotic treatment in children and adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-18 years (at any point during study participation
* BMI > 85th percentile
* One or more DSM-IV diagnoses, including disruptive behavior disorders (attention deficit disorder, conduct disorder, oppositional defiant disorder and disruptive behavior disorder not otherwise specified), affective disorders (bipolar affective disorder, major depressive disorder and mood disorder not otherwise specified), anxiety disorders (generalized anxiety disorder, obsessive compulsive disorder, separation anxiety, social and other specific phobias) as well as other disorders, including autism spectrum disorders (autistic disorder, Asperger's Syndrome and pervasive developmental disorder not otherwise specified), psychotic disorders (schizophreniform disorder, schizophrenia and psychotic disorder not otherwise specified) and movement disorders (tic disorder, Tourette's Syndrome)
* At least 12 weeks of treatment and no more than approximately 12 months treatment with risperidone or olanzapine immediately prior to study enrollment (assuming that the initial phase of prior treatment involved a dose titration; clinically minor dosing deviations such as changes in dose or missed doses will be evaluated for inclusion by the PI on an individual basis)
* No clinically significant changes in permitted medications (e.g., stimulants) for 1 month prior to Baseline Evaluations (inclusion determined by evaluation on an individual basis by the PI)
* Clinically significant weight gain during an initial course of antipsychotic treatment; for non-MEAC participants, this is defined as > 10% increase from baseline weight during the prior treatment if treatment lasted approximately 5-12 months or defined as > 7% increase from baseline weight during the prior treatment if treatment lasted approximately 3-4 months (based on the totality of information from primary care provider, school and home); for prior MEAC participants, clinically significant weight gain is defined as > 7% increase from baseline weight over the course of the 3 month MEAC study and/or > 10% increase in total body fat as measured by DEXA during the MEAC study
* Score of > 18 on the irritability subscale of the Aberrant Behavior Checklist prior to initiating antipsychotic treatment: MEAC participants will automatically meet this criterion based on similar inclusion criteria for MEAC; for non-MEAC participants, the ABC questionnaire will be administered to parents and one or more collateral source (such as a teacher, social worker or alternate caregiver) by study staff to retrospectively gather information about symptoms of irritability and aggression prior to initiation of antipsychotic treatment. Non-MEAC participants with a retrospective, consensus (i.e., clinician evaluation of all available sources of ABC data) ABC irritability subscale score of > 18 in proximity to (e.g., within 3 months of) initiation of treatment will be included (based on combined evaluation of the totality of available corroborative resources), and viii) Clinically significant improvement in psychiatric symptoms during the initial course of antipsychotic based on > 30% decrease in ABC irritability score from baseline to endpoint in the MEAC study or a retrospective consensus of 30% decrease in ABC over the prior course of treatment OR a CGI-I score of 2 or better or psychiatric symptoms experienced for at least 1 month prior to enrollment as measured by a CGI-S score of 3 or less (mildly ill).

Exclusion Criteria:

* Active suicidality
* The presence of any serious medical disorder or condition that may, in the judgment of the PI, confound the assessment of relevant biologic measures or diagnoses, including: clinically significant organ system dysfunction; significant endocrine disease, including diabetes mellitus; coagulopathy; significant anemia; or significant acute infection; or pregnancy
* Participants taking within the last 3 months any glucose lowering agent, lipid lowering agent, exogenous testosterone, recombinant human growth hormone, or any other endocrine agent that might confound substrate metabolism, oral glucocorticoids (glucocorticoid nasal spray and inhalers are permitted), sedating antihistamines (non-sedating antihistamines like Claritin (loratadine) and Zyrtec (cetirizine) are permitted), non- serotonin selective reuptake inhibitor antidepressants and mood stabilizing agents (exposure to SSRI's, stimulants, clonidine and guanfacine permitted)
* IQ < 70 (based on school records and/or evaluation by clinician)
* Current substance abuse; vi) past history of, or current dyskinesia
* Stimulant dosage higher than approximately 2 mg/kg/day methylphenidate or equivalent dose of non-methylphenidate stimulant
* Participants who at baseline have elevated total cholesterol or low density lipoprotein cholesterol (> 95th percentile for age and gender) will be excluded based on recent American Academy of Pediatric recommendations to treat this level of dyslipidemia with pharmacotherapy,(63) unless is can be documented that they achieved the > 95th percentile dyslipidemia during antipsychotic treatment but did not have it at baseline (e.g., MEAC recruits) given the clinical equipoise around whether the planned intervention could lower lipids back below the threshold and allow them to avoid the risks of lipid lowering drugs
* Baseline fasting triglyceride > 400 mg/dl

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2009-11; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
Changes in per cent of body fat | 16 weeks

SECONDARY OUTCOMES:
Changes in insulin sensitivity | 16 weeks
Psychiatric safety and tolerability | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John W Newcomer, MD, Principal Investigator — Washington University School of Medicine and Florida Atlantic University